CLINICAL TRIAL: NCT01004601
Title: Chang Gung Memorial Hospital, Chang Gung University, College of Medicine, Taipei, Taiwan
Brief Title: Low Dose Weekly Docetaxel Versus Pemetrexed in Previously Treated Advanced Non-Small-Cell Lung Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Chang Gung Memorial Hospital, Chang Gung Memorial Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 98-2587B
Record Dates: First submitted 2009-10-27; First posted 2009-10-30 (Estimated); Last update posted 2009-10-30 (Estimated); Status verified 2009-10

CONDITIONS: Non Small Cell Lung Cancer
Keywords: pretreated failure advanced stage IIIb/IV NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Docetaxel; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- low dose docetaxel (Active Comparator): Low dose single docetaxel (30 mg/m2 on days 1 and 8 every 3 weeks)
  Interventions: Drug: docetaxel
- Pemetrexed (Active Comparator): Pemetrexed (500 mg/m2 every 3 weeks)
  Interventions: Drug: pemetrexed

INTERVENTIONS:
Drug: docetaxel — patients at one university-affiliated hospital received low dose single docetaxel (30 mg/m2 on days 1 and 8 every 3 weeks)following failure of previous treatment stage IIIb/IV NSCLC.
  Arms: low dose docetaxel
Drug: pemetrexed — patients at one university-affiliated hospital received pemetrexed (500 mg/m2 every 3 weeks) following failure of previous treatment stage IIIb/IV NSCLC.
  Arms: Pemetrexed

SUMMARY:
Docetaxel and pemetrexed have been validated for previously treated advanced non-small cell lung cancer (NSCLC); however, tolerability is a concern with the docetaxel (tri-weekly 75 mg/m2 schedule). The investigators conducted this study to compare the efficacy and toxicity of weekly low-dose docetaxel versus tri-weekly pemetrexed for previously treated advanced NSCLC.

DETAILED DESCRIPTION:
We have been following a schedule of weekly low dose docetaxel (30 mg/m2 on days 1 and 8 every 3 weeks; 60 mg/m2 accumulated dose for each cycle) at our hospital in an effort to achieve better tolerability. We therefore performed an exploratory study, by statistical analyses, to investigate the efficacy and toxicity of such a low dose docetaxel schedule compared to that of pemetrexed in patients with NSCLC who have failed previous chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* stage IIIb or IV NSCLC
* previous treatment with chemotherapy or tyrosin kinase inhibitor
* performance status less than 2

Exclusion Criteria:

* age less 18 years
* pregnancy
* performance status 3-4

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2005-03; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Objective response rate | at least 3 cycles

SECONDARY OUTCOMES:
PFS-progression free survival | the time from the first cycle of chemotherapy to documented progression, or death from any cause
OS-overall survival | from the start date of the treatment to death or to the last follow-up visit

CONTACTS AND LOCATIONS:
Overall Officials: Han-Pin Kuo, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taipei, Taipei, Taiwan

REFERENCES:
- [Background] Hanna N, Shepherd FA, Fossella FV, Pereira JR, De Marinis F, von Pawel J, Gatzemeier U, Tsao TC, Pless M, Muller T, Lim HL, Desch C, Szondy K, Gervais R, Shaharyar, Manegold C, Paul S, Paoletti P, Einhorn L, Bunn PA Jr. Randomized phase III trial of pemetrexed versus docetaxel in patients with non-small-cell lung cancer previously treated with chemotherapy. J Clin Oncol. 2004 May 1;22(9):1589-97. doi: 10.1200/JCO.2004.08.163. PMID 15117980
- [Background] Di Maio M, Perrone F, Chiodini P, Gallo C, Camps C, Schuette W, Quoix E, Tsai CM, Gridelli C. Individual patient data meta-analysis of docetaxel administered once every 3 weeks compared with once every week second-line treatment of advanced non-small-cell lung cancer. J Clin Oncol. 2007 Apr 10;25(11):1377-82. doi: 10.1200/JCO.2006.09.8251. PMID 17416857
- [Background] Schuette W, Nagel S, Blankenburg T, Lautenschlaeger C, Hans K, Schmidt EW, Dittrich I, Schweisfurth H, von Weikersthal LF, Raghavachar A, Reissig A, Serke M. Phase III study of second-line chemotherapy for advanced non-small-cell lung cancer with weekly compared with 3-weekly docetaxel. J Clin Oncol. 2005 Nov 20;23(33):8389-95. doi: 10.1200/JCO.2005.02.3739. PMID 16293869
- [Background] Kunitoh H, Watanabe K, Onoshi T, Furuse K, Niitani H, Taguchi T. Phase II trial of docetaxel in previously untreated advanced non-small-cell lung cancer: a Japanese cooperative study. J Clin Oncol. 1996 May;14(5):1649-55. doi: 10.1200/JCO.1996.14.5.1649. PMID 8622084
- [Background] Scagliotti GV, Parikh P, von Pawel J, Biesma B, Vansteenkiste J, Manegold C, Serwatowski P, Gatzemeier U, Digumarti R, Zukin M, Lee JS, Mellemgaard A, Park K, Patil S, Rolski J, Goksel T, de Marinis F, Simms L, Sugarman KP, Gandara D. Phase III study comparing cisplatin plus gemcitabine with cisplatin plus pemetrexed in chemotherapy-naive patients with advanced-stage non-small-cell lung cancer. J Clin Oncol. 2008 Jul 20;26(21):3543-51. doi: 10.1200/JCO.2007.15.0375. Epub 2008 May 27. PMID 18506025
- [Background] Weiss GJ, Langer C, Rosell R, Hanna N, Shepherd F, Einhorn LH, Nguyen B, Paul S, McAndrews P, Bunn PA Jr, Kelly K. Elderly patients benefit from second-line cytotoxic chemotherapy: a subset analysis of a randomized phase III trial of pemetrexed compared with docetaxel in patients with previously treated advanced non-small-cell lung cancer. J Clin Oncol. 2006 Sep 20;24(27):4405-11. doi: 10.1200/JCO.2006.06.7835. PMID 16983108
- [Background] Chen YM, Shih JF, Perng RP, Tsai CM, Whang-Peng J. A randomized trial of different docetaxel schedules in non-small cell lung cancer patients who failed previous platinum-based chemotherapy. Chest. 2006 Apr;129(4):1031-8. doi: 10.1378/chest.129.4.1031. PMID 16608954
- [Background] Bria E, Cuppone F, Ciccarese M, Nistico C, Facciolo F, Milella M, Izzo F, Terzoli E, Cognetti F, Giannarelli D. Weekly docetaxel as second line chemotherapy for advanced non-small-cell lung cancer: meta-analysis of randomized trials. Cancer Treat Rev. 2006 Dec;32(8):583-7. doi: 10.1016/j.ctrv.2006.07.003. Epub 2006 Aug 21. PMID 16919884